CLINICAL TRIAL: NCT03885843
Title: A Prospective, Multicenter, Blind, Randomized and Controlled Trial of Selected Renal Denervation by Renal Nerve Mapping for the Treatment of Hypertension (HTN) in the Absence of Antihypertensive Medications (OFF MED)
Brief Title: Sympathetic Mapping/ Ablation of Renal Nerves Trial (SMART) HTN-OFF MED Study
Acronym: SMART OFF-MED
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Second Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Yuehui Yin, Director of the Department, The Second Affiliated Hospital of Chongqing Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SMART HTN-OFF MED
Record Dates: First submitted 2019-03-20; First posted 2019-03-22 (Actual); Last update posted 2019-03-25 (Actual); Status verified 2019-03

CONDITIONS: Essential Hypertension; Vascular Diseases; Cardiovascular Diseases
MeSH Terms: conditions — Essential Hypertension; Vascular Diseases; Cardiovascular Diseases | interventions — Denervation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RDN Group (Experimental): renal nerve stimulation, mapping and denervation using the SyMapCath I™ Catheter and SYMPIONEER S1™ Stimulator/Generator after renal angiography.
  Interventions: Procedure: Renal nerve stimulation, mapping and denervation
- Sham Group (Sham Comparator): renal artery angiography group, without any renal nerve stimulation, mapping or denervation
  Interventions: Procedure: Sham Procedure: Renal angiography

INTERVENTIONS:
Procedure: Renal nerve stimulation, mapping and denervation — After a renal angiography according to standard procedures, subjects remain blinded and are immediately treated with the renal nerve stimulation, mapping and denervation procedure after randomization.
  Arms: RDN Group
Procedure: Sham Procedure: Renal angiography — After a renal angiography according to standard procedures, subjects remain blinded and remain on the catheterization lab table for at least 20 minutes prior to introducer sheath removal
  Arms: Sham Group

SUMMARY:
To evaluate the efficacy and safety of selected renal sympathetic denervation using SyMapCath I™ Catheter and SYMPIONEER S1™ Stimulator/Generator in patients with hypertension in the absence of antihypertensive medications, or till the negative result was given by urinary antihypertensive drugs detection of high-performance liquid chromatography-tandem mass spectrometry (HPLC-MS/MS) after at least two weeks of drug elution period.

Then Office systolic blood pressure (SBP) is still ≥ 150mmHg, < 180mmHg, diastolic blood pressure (DBP) ≥ 90mmHg, and 24-hour mean SBP of ambulatory blood pressure measurement (ABPM) is ≥130mmHg, or day-time mean SBP ≥135mmHg, or night-time mean SBP ≥120mmHg, and all SBP of ABMP record <170mmHg.

After then the patient will be included when the results of bilateral renal angiography meet the requirements of renal nerve stimulation, mapping and denervation conditions.

DETAILED DESCRIPTION:
This is a prospective, multicenter, blind, randomized and controlled trial, in which patients are of essential hypertension, but in the absence of antihypertensive medications. The patients will be informed, consent and get into a screening process. After at least two weeks of drug elution period HPLC-MS/MS urinary antihypertensive drugs detection will be given till the negative result, or one extra week of drug elution period will be given for the second urinary drugs analysis. Then Office systolic blood pressure (SBP) is still ≥ 150mmHg, < 180mmHg, diastolic blood pressure (DBP) ≥ 90mmHg, and 24-hour mean SBP of ambulatory blood pressure measurement (ABPM) is ≥130mmHg, or day-time mean SBP ≥135mmHg, or night-time mean SBP ≥120mmHg, and all SBP of ABMP record <170mmHg.

These patients will conduct renal angiography, and the meet inclusion criteria individuals will be allocated to either renal nerve stimulation, mapping and denervation group (RDN group) or renal artery angiography group (Sham group) by a randomizing system in a 1:1 ratio (80 patients, 40 pairs). Physicians who perform post-procedure patient management and physicians who perform renal denervation procedures are blinded to each other.

Patients will be followed at the 2nd day, the 7th day after the procedure or at discharge from hospital, 1st month, 2nd month, 3rd month. Urine samples will be collected for drug tests to determine drug compliance of a patient.

Data collecting/management/statistical analysis and laboratory tests will be performed by independent, qualified organizations. Independent Data Safety and Monitoring Board/Clinical Events Committee (DSMB/CEC) are formed and responsible for assessments of protocol deviations and natures of serious adverse events (SAEs).

ELIGIBILITY:
Inclusion Criteria:

1. Male and non-pregnant female subjects, 18≤age≤65
2. Essential hypertension
3. Office SBP ≥150mmHg and < 180mmHg; and DBP ≥90mmHg
4. Average 24-hour ABPM systolic blood pressure is ≥130mmHg, or day-time mean SBP ≥135mmHg, or night-time mean SBP ≥120mmHg, and all SBP of ABMP record <170mmHg
5. HPLC-MS/MS urinary antihypertensive drugs detection shows negative result after at least two weeks of drug elution period, or one extra week of drug elution period will be given for the second urinary drugs analysis; and the urinary drugs detection can be given in screening date for the subjects without antihypertensive history
6. Renal arteries meet the criteria of renal nerve stimulation, mapping and denervation; and at least one positive-response point occurs in each renal artery
7. Patient understands the purpose of this study, and is willing to participate and sign the Informed Consent
8. Patient is compliant and willing to complete clinical follow-up.

Exclusion Criteria:

1. Renal artery anatomy is unqualified including：

1. Diameter <3.5mm or treatable length <25mm;
2. Multiple renal arteries and the main renal artery supplies a fraction of the blood flow less than 75%
3. Renal artery stenosis >50% or any renal artery aneurysms on either side
4. History of renal artery percutaneous transluminal angioplasty (PTA), including balloon angioplasty and stenting 2. eGFR <45ml/min/1.73m2 (MDRD formula) 3. Hospitalized within one year due to hypertensive crisis 4. Pulse pressure>80mmHg, or isolated systolic hypertension 5. During running in period, using any antihypertensive drugs without prescription and urinary drugs test shows positive.

6. Participated other clinical trials including both drug and medical device studies within 3 months enrollment 7. Female with pregnant or lactating, or having plans for pregnancy within 1 year 8. Patient with sleep apnea who needs chronic oxygen-breathing or mechanical ventilation support (for example, tracheostomy) 9. Patients previously or currently suffering from following diseases:

1. Essential pulmonary arterial hypertension
2. Type I diabetes
3. Severe cardiac valvular stenosis with contradictions to significantly reduce blood pressure
4. History of myocardial infraction (MI), unstable angina, syncope or cerebrovascular accidents within half year.
5. History of primary aldosteronism, pheochromocytoma, aorta stenosis, hyperthyroidism or hyperparathyroidism
6. Any disease conditions interfering the measurement of blood pressure (for instance, severe peripheral artery diseases, abdominal artery aneurysm, hemorrhagic disorders such as thrombocytopenia, hemophilia and severe anemia)
7. Plans to have surgery or cardiovascular interventions within following 6 months
8. Alcohol abuse or unknown drug dependence history
9. Neuroticisms such as depression or anxiety disorders
10. Non-compliant patients unable to finish the research per physician's requests 10. There is no positive-response point in any renal artery, or any contradictions to conduct renal artery stimulation and ablation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-06-01 (Estimated); Primary Completion 2020-01-01 (Estimated); Study Completion 2020-04-01 (Estimated)

PRIMARY OUTCOMES:
Change in office systolic blood pressure | 3 months after the treatment

SECONDARY OUTCOMES:
Change in average 24-hour Ambulatory Blood Pressure Monitoring (ABPM) systolic blood pressure (SBP) | 3 months
Change in average day-time ABPM SBP | 3 months
Change in average night-time ABPM SBP | 3 months
Change in office diastolic blood pressure (DBP) | 3 months
Change in mean arterial blood pressure | 3 months
Change in the blood catecholamines levels of pre-procedure and 3 months after the procedure | 3 months
Rate of renal artery stenosis assessed by CT angiography | 3 months
  (stenosis > 70% )
Rate of severe renal dysfunction | 3 months
  eGFR<15ml/min/m2 or renal function replacement therapy needed
Rate of adverse events (AEs), SAEs, and severe cardio-cerebrovascular events | 3 months
Rate of all-cause death | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- 2ndChongqingMU, Chongqing, Chongqing Municipality, China